CLINICAL TRIAL: NCT00456105
Title: Early Post-Operative Dysglycemia in Patients With and Without Diabetes Post-Infrainguinal Bypass Surgery and the Effectiveness of a Diabetes Action Team in the Management of Diabetes Post Infrainguinal Bypass Surgery on Glycemic Control, Length of Stay, and Infection Rates: A Pilot Study
Brief Title: The Effect of a Diabetes Action Team in Patients Post Infrainguinal Bypass Surgery With and Without Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped due to lack of resources of the study coordinator's time
Sponsor: University of British Columbia (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Graydon Meneilly, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H05-70482
Record Dates: First submitted 2007-04-02; First posted 2007-04-04 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Type 2 Diabetes; Peripheral Vascular Disease
Keywords: Type 2 diabetes; Post-op dysglycemia; Peripheral vascular disease; Infrainguinal bypass surgery
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Subjects with diabetes who plan to undergo elective infrainguinal bypass surgery will receive standard diabetes care by their admitting physician, post operatively until hospital discharge and post discharge in the community.
  Interventions: Behavioral: Subjects with diabetes who plan to undergo elective infrainguinal bypass surgery will receive standard diabetes care by their admitting physician
- 2 (Experimental): Subjects with diabetes who plan to undergo elective infrainguinal bypass surgery will receive diabetes care under the direction of the Diabetes Action Team post operatively until hospital discharge and post discharge in the community. The Diabetes Action team will consist of a nurse coordinator who is a Certified Diabetes Educator (CDE) and a team of physicians specialized in the management of diabetes.
  Interventions: Behavioral: Subjects with diabetes who plan to undergo elective infrainguinal bypass surgery will receive diabetes care under the direction of the Diabetes Action Team
- 3 (Placebo Comparator): Subjects without diabetes will have their blood glucose levels monitored while in the hospital.
  Interventions: Behavioral: Subjects without diabetes will have their blood glucose levels monitored while in the hospital

INTERVENTIONS:
Behavioral: Subjects with diabetes who plan to undergo elective infrainguinal bypass surgery will receive standard diabetes care by their admitting physician — See Detailed Description.
  Arms: 1
Behavioral: Subjects with diabetes who plan to undergo elective infrainguinal bypass surgery will receive diabetes care under the direction of the Diabetes Action Team — See detailed description.
  Arms: 2
Behavioral: Subjects without diabetes will have their blood glucose levels monitored while in the hospital — See detailed description.
  Arms: 3

SUMMARY:
Diabetes is a very common illness. Approximately 4% of British Columbians have diabetes. However, at least 20% of people admitted to acute care hospitals have diabetes. People with diabetes are at a higher risk for developing complications after surgery including infection and prolonged hospital stay, especially if blood sugars are high.

The researchers are testing a Diabetes Action Team to see if their involvement in patient care after surgery improves blood glucose control, duration of stay in hospital, and infection rates.

DETAILED DESCRIPTION:
This trial will randomize subjects with diabetes who plan to undergo elective infrainguinal bypass surgery to receive either standard diabetes care by their admitting physician, or diabetes care under the direction of the Diabetes Action Team post operatively until hospital discharge and post discharge in the community. Subjects without diabetes will have their blood glucose levels monitored while in the hospital. The Diabetes Action team will consist of a nurse coordinator who is a Certified Diabetes Educator (CDE) and a team of physicians specialized in the management of diabetes. The study will not increase the length of the hospital stay.

ELIGIBILITY:
Inclusion Criteria:

Non-Diabetes:

* Fasting blood glucose < 7.0 mmol/L or a random blood glucose of < 11.1 mmol/L

Diabetes:

* Poorly controlled type 2 diabetes (fasting plasma glucose greater than or equal to 7.0 or random plasma glucose greater than or equal to 10.0 mmol/L)
* Newly diagnosed type 2 diabetes (fasting plasma glucose greater than or equal to 7.0 mmol/L or random plasma glucose greater than or equal to 11.1 mmol/L)
* Age > 30
* English-speaking
* Agrees to participate in the study and lives in the Lower Mainland

Exclusion Criteria:

* Scheduled to undergo surgery other than infrainguinal bypass surgery
* Under 30 years of age
* Living outside of Lower Mainland
* Cannot speak and understand English

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Glycemic control

SECONDARY OUTCOMES:
Length of stay
Infection
Readmission

CONTACTS AND LOCATIONS:
Overall Officials: Graydon Meneilly, MD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia Gerontology & Diabetes Research Centre, Vancouver, British Columbia, Canada